CLINICAL TRIAL: NCT04817943
Title: Comparison of Esophageal and Tracheal Temperature in the Patients Using Breathing Circuit With Heated Wire Humidifier
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2021-028
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: The Patients Who Underwent General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non applicable — When the patient enters the operating room, oxygen saturation, blood pressure, and electrocardiogram are monitored, and general anesthesia is induced using 1-2 mg/kg of 1% propofol. 0.8 mg/kg of rocuronium, a neuromuscular blocker, is injected intravenously, and a human endotracheal tube is intubated. A thermometer is attached to the inside of the double-layered endotracheal tube cuff, which measures the temperature in the trachea. After the endotracheal intubation is performed, the esophageal thermometer is inserted, and from this point, the temperature measured by the esophageal thermometer and the thermometer of the endotracheal tube are recorded. The temperature immediately after insertion of the esophageal thermometer is set as Tbaseline, and the temperature of the esophagus and trachea, the temperature of the operating room, and the temperature of breathing circuit with heated wire humidifier are recorded every 5 minutes from thereafter until the end of the operation.

SUMMARY:
When using a breathing circuit with heated wire humidifier, investigators will check if the temperature measured by the thermometer of the endotracheal tube is more than 0.25 degrees apart from the temperature measured by the esophageal thermometer. Through this, in the case of patients who need to use a breathing circuit with heated wire humidifier, investigators will find out whether it is appropriate to use an esophageal or endotracheal thermometer.

DETAILED DESCRIPTION:
It is known that hypothermia occurs in approximately 50-90% of surgical patients under general anesthesia, and intraoperative hypothermia can lead to various complications such as wound infection, coagulation disorders, increased frequency of cardiac complications, ventricular fibrillation, prolonged effects of anesthesia drugs, shivering, and weakened immune function. Additionally, inadequate maintenance of temperature during surgery can result in delayed discharge from the recovery room, delayed recovery, and extended hospitalization. Therefore, accurate measurement of body temperature and active temperature management are crucial during surgery. Although there are various sites for temperature measurement, measuring the core body temperature in well-perfused deep tissues, which have a higher temperature and greater reliability than other sites, is essential. While esophageal temperature measurement is commonly used in patients undergoing general anesthesia, there may be cases where esophageal temperature probe cannot be inserted due to bleeding tendencies or lesions in the esophagus. In such cases, measuring temperature through the tympanic membrane or an endotracheal device becomes possible, but using a heated humidification breathing circuit for patient warming may affect the endotracheal temperature. Although there are animal study results comparing esophageal temperature and endotracheal temperature, research on the comparison of esophageal and endotracheal temperatures in humans is limited, and there is no study on the comparison of esophageal and endotracheal temperatures when using a heated humidification breathing circuit. The investigators aim to verify whether there is a temperature difference of 0.25 degrees or more between the temperature measured through the endotracheal device and the temperature measured by the esophageal thermometer when using a heated humidification breathing circuit. Through this investigation, they seek to determine which thermometer, either esophageal or endotracheal, is more appropriate to use in patients requiring the use of a heated humidification breathing circuit.

ELIGIBILITY:
Inclusion Criteria:

* males and females between the ages of 20 and 60 and meet the criteria for classification I and II of the American Society of Anesthesiology

Exclusion Criteria:

* Patients with a predisposition for bleeding
* Patients with a history of inability to insert an esophageal thermometer (esophageal varices, esophageal stenosis, esophageal malformation, and anatomical deformation after esophageal surgery)
* pregnant woman

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Among the patients undergoing surgery that requires more than 2 hours of general anesthesia and the use of a breathing circuit with heated wire humidifier
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Esophageal and tracheal temperature measurement | during operation
  Esophageal and tracheal temperature measurement in patients undergoing surgery that requires more than 2 hours of general anesthesia and the use of breathing circuit with heated wire humidifier

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Department of Anesthesia and Pain Medicine, School of Medicine, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea